CLINICAL TRIAL: NCT02183649
Title: A Phase I, Single-dose, Two-way Crossover Study to Investigate Tolerability and Potential ECG Effects After a Single Oral Dose of 192 mg Pentoxyverine Citrate (Corresponding to 121.5 mg Pentoxyverine Base) in Healthy Male and Female Volunteers (Randomised, Single-blind, Placebo-controlled)
Brief Title: Tolerability and Potential ECG Effects After a Single Oral Dose of Pentoxyverine Citrate in Healthy Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1265.1
Record Dates: First submitted 2014-07-07; First posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
MeSH Terms: interventions — carbetapentane

STUDY DESIGN:
Who Masked: Participant

ARMS (1):
- pentoxyverine citrate vs. placebo (Experimental): All subjects were allocated to receive both verum and placebo in randomised order
  Interventions: Drug: pentoxyverine citrate; Drug: Placebo

INTERVENTIONS:
Drug: pentoxyverine citrate
Drug: Placebo

SUMMARY:
The primary objective of this trial was to investigate the potential effects of pentoxyverine on the ECGs of healthy subjects. A secondary objective was the exploration of safety and tolerability. Pharmacokinetics (PK) were only to be investigated if necessary for the explanation of ECG effects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female subjects according to the following criteria:

   Based upon a complete medical history, including the physical examination, vital signs (blood pressure (BP), pulse rate (PR)) 12-lead ECG, clinical laboratory tests
2. Age ≥21 and ≤45 years
3. Body Mass Index (BMI) ≥18.5 and ≤29.9 kg/m²
4. Signed and dated written informed consent prior to admission to the study in accordance with GCP and the local legislation.

Exclusion Criteria:

1. Any finding of the medical examination (including BP, PR, and ECG) deviating from normal and of clinical relevance
2. Any evidence of a clinically relevant concomitant disease
3. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
4. Surgery of the gastrointestinal tract (except appendectomy)
5. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
6. History of relevant orthostatic hypotension, fainting spells or blackouts.
7. Chronic or relevant acute infections
8. History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
9. Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
10. Use of drugs which might reasonably influence the results of the trial or that prolong the QT/QTc interval based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
11. Participation in another trial with an investigational drug within two months prior to administration or during the trial
12. Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
13. Inability to refrain from smoking on trial days
14. Alcohol abuse (more than 60 g/day)
15. Drug abuse
16. Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
17. Excessive physical activities (within one week prior to administration or during the trial)
18. Any laboratory value outside the reference range that is of clinical relevance
19. Inability to comply with dietary regimen of trial site
20. A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 ms);
21. A history of additional risk factors for torsade de pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2009-11; Primary Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
changes from baseline in QTc interval | up to 24 hours

SECONDARY OUTCOMES:
number of adverse events | up to day 44
Blood pressure change from baseline | up to day 44
Pulse rate change from baseline | up to day 44
assessment of global tolerability by 4-point scale | up to day 44